CLINICAL TRIAL: NCT04573166
Title: Personalized Atrial Septostomy With Combined Use of Radiofrequency-ablation and Balloon-dilation: First-in-human Study in Heart Failure
Brief Title: Personalized Atrial Septostomy for Heart Failure
Acronym: PAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-8
Record Dates: First submitted 2020-09-20; First posted 2020-10-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Heart Failure, Diastolic
Keywords: Heart failure; atrial septostomy
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: After left and right catheterization, CURB procedure will be performed in all patients. The first step is RFA on fossae ovalis; and then graded BAS is carried out after transseptal puncture; finally, RFA is repeated around the fenestration-rim created with BAS. The fenestration-size will be determined based on the levels of AOP and MLAP, and the immediate size of fenestration will be evaluated with intra-cardiac echocardiography. The patency and size of fenestration will be followed up for 12 months. During the period of follow up, the other evaluations will include the improvement in exercise tolerance, major adverse cardiac and/or cerebrovascular events (MACCE), reduction of PAWP/MLAP at rest, cardiac remodeling, myocardial injury, and so on.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CURB procedure (Experimental): Personalized atrial septostomy with combined use of radiofrequency-ablation and balloon-dilation (CURB)
  Interventions: Procedure: Personalized atrial septostomy with combined use of radiofrequency-ablation and balloon-dilation

INTERVENTIONS:
Procedure: Personalized atrial septostomy with combined use of radiofrequency-ablation and balloon-dilation — After left and right catheterization, CURB procedure will be performed in all patients. The first step is RFA on fossae ovalis; and then graded BAS is carried out after transseptal puncture; finally, RFA is repeated around the fenestration-rim created with BAS. The fenestration-size will be determined based on the level of MLAP, and the immediate size of fenestration will be evaluated with intra-cardiac echocardiography. The patency and size of fenestration will be followed up for 6 months. During the period of follow up, the other evaluations will include the improvement in exercise tolerance, major adverse cardiac and/or cerebrovascular events (MACCE), reduction of PAWP/MLAP at rest, cardiac remodeling, myocardial injury, and so on.

SUMMARY:
This study aims to investigate the safety and efficacy of personalized atrial septostomy (PAS) with combined use of radiofrequency-ablation and balloon-dilation (CURB) in heart failure with reduced ejection fraction (HFrEF) and heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Atrial septostomy is an important palliative therapy in heart failure with reduced ejection fraction (HFrEF) and heart failure with preserved ejection fraction (HFpEF) . Though the safety of balloon atrial septostomy (BAS) is satisfactory, the incidence of spontaneous closure is higher, which limits the clinical utilization of this procedure. The device-implantation improves the long-term patency. However, the created fenestration is limited with fixed size and it is further complicated with the potential device-related complications.

Radiofrequency catheter ablation (RFA) has the potential to cause irreversible damage around the rim of fenestration created with BAS, which might prevent the re-adhesion of the septal remnants. In addition, RFA on fossae ovalis might reduce the elastic recoil of local tissue and contribute to create larger inter-atrial fenestration with same BAS procedure. Therefore, the combined use of radiofrequency-ablation and balloon-dilation (CURB) might become a novel procedure to create a stable inter-atrial fenestration.

In this study, the adult patients who have HFrEF and HFpEF refractory to medical therapy may be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Symptomatic heart failure in NYHA class III or IV ambulatory;
3. Optimal medical therapy of heart failure according to European Society of Cardiology (ESC) guidelines for last 6 months;
4. LVEF ≥ 45%;
5. Elevated left heart filling pressures: left ventricular end-diastolic pressure (LVEDP) or pulmonary capillary wedge pressure (PCWP) ≥ 18 mmHg at rest;
6. LVEDP or PCWP-Mean right atrial pressure (MRAP) ≥ 5 mmHg;
7. Systolic blood pressure ≥ 90 mmHg.

Exclusion Criteria:

1. Acute infection or sepsis;
2. Intra-cardiac mass, thrombus or vegetation;
3. Evidence of right heart failure (TAPSE < 14 mm);
4. Pulmonary hypertension (PASP > 60 mmHg);
5. Associated atrial septal defect or large patent foramen ovale with significant left to right shunt in rest;
6. TIA or stroke within the last 6 months;
7. Thromboembolic events within the last 6 months;
8. Hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy as cause of heart failure;
9. Valvular diseases requiring therapy according to current ESC guidelines;
10. Life expectancy < 1 year for non-cardiovascular reasons.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical change | 12 months
  Distance in 6 minutes walk test
The size of created-fenestration | 12 months
  The change of created-fenestration size evaluated with echocardiography

SECONDARY OUTCOMES:
The percent of subjects who experience major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  Peri-procedural, and 12 months MACCE and systemic embolic events in patients after CURB procedure.
Change of PAWP or MLAP at rest | 12 months
  Pulmonary capillary wedge pressure (PCWP)/MLAP at rest evaluated with right heart catheterization
Change of cardiac remodeling | 12 months
  The change in cardiac chamber and function evaluated with MSCT and CMR
Myocardial remodeling | 12 months
  The myocardial molecular imaging evaluated with PET-CT

CONTACTS AND LOCATIONS:
Overall Officials: Chaowu Yan, PhD and MD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (2):
- China (2):
  - National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences,Fuwai Hospital, Beijing, Beijing Municipality
  - Yan Chaowu, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan C, Li H, Wan L, Liu A, Yundan P, Guo T, Hua L, Wang L, Fang W. Left atrial pressure normalisation by graded radiofrequency atrial septostomy in heart failure with preserved ejection fraction: a single-arm pilot study. Heart. 2025 Oct 14;111(21):1020-1027. doi: 10.1136/heartjnl-2025-325929. PMID 40425275